CLINICAL TRIAL: NCT04441476
Title: Ethical and Psychological Support for Health Care Professions in Intensive Care Units in the COVID19 Pandemic Context: Adequacy With Needs and Psychological Impact Crisis and Post-crisis
Acronym: PsyCOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUENOT SERI 2020
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-06

CONDITIONS: Psychological Strain
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU staff
  Interventions: Other: Questionnaires; Other: psychological and sociological interviews

INTERVENTIONS:
Other: Questionnaires — An online questionnaire (Limesurvey platform) will be made available at 4 different times (M0, M1, M2 and M6).
  * The first questionnaires (M0 and M1) will include a component for professional characterization. Generic and specific stress factors related to ICU and the current pandemic and collective and individual defensive strategies will also be collected in M0 and M1.
  * At M2 and M6, the traumatic impact of the crisis, burnout, signs of depression and recourse to internal or external support in the department (occupational medicine, support unit) will be collected.
Other: psychological and sociological interviews — conducting semi-directive psychological interviews (40 interviews in M2, 40 interviews in M6).
  sociological interviews: 40 (20 in M1-M2 then 20 in M6) in order to understand the consequences of the epidemic on daily life, both intra-family and micro-social.

SUMMARY:
The intensive care unit occupies a particular place in our health care system. The urgency of the clinical situations, the proportion of deaths encountered, and the daily workload is likely to generate suffering among staff. The health crisis linked to SARS-COV-2 is unprecedented and has leads to the unprecedented mobilisation of care providers, particularly in the ICU. Faced with the massive and growing influx of patients, human, therapeutic and material resources are overwhelmed and the teams are faced with an unusually heavy workload in a context of extreme tension. These professionals are thus exposed to a risk of over-investment, in a context of acute and repetitive stress, over an indeterminate period of time combining workload, emotional intensity with specific ethical issues, simultaneously affecting the professional sphere but also the personal and family sphere (confinement, risk of contamination). Now more than ever, the mental health of caregivers is an important concern, as highlighted by the CCNE. Mental health is understood in the way in which the individual responds specifically to work-related suffering by developing individual and collective defensive strategies. Thus, the issue of mental health in the ICU cannot be considered without taking into account the strategies that professionals put in place to combat stress and to contribute or not to the construction and stabilization of the work collective (collaboration, support). Ethical and/or psychological support systems have been set up in most of the establishments involved in the care of Covid-19 patients. However, the adequacy of these systems relative to the needs of professionals during and after the crisis is not yet known. We hypothesize that the psychological and social repercussions of this pandemic as well as the individual and collective strategies deployed by ICU care providers to deal with it will evolve in view of the progression of the crisis but also of the various types of support, particularly psychological and/or ethical, available to them.

ELIGIBILITY:
Inclusion Criteria:

* The study population is the entire ICU staff of the participating centres, whether they are permanently or transiently assigned to these units and/or the institution, whether they are students or not.

Professionals involved in psychological and ethical support structures may also be interviewed to provide the information necessary to describe and evaluate the organisations and their evolution.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nursing staff in French hospitals
Sampling Method: Probability Sample
Enrollment: 3080 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
PS-ICU Scale Score | Through study completion, an average of 6 months after the epidemic peak
  This scale integrates generic stressors as well as factors specific to intensive care and crises.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France